CLINICAL TRIAL: NCT02571205
Title: Observational Study of Clinical Outcomes for Testosterone Treatment of Pubertal Delay in Duchenne Muscular Dystrophy
Brief Title: Testosterone Therapy for Pubertal Delay in Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-003195-68
Record Dates: First submitted 2015-08-24; First posted 2015-10-08 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: testosterone; pubertal delay
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Puberty, Delayed | interventions — Testosterone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples to be collected as part of Biobank
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sustanon (testosterone) — Standard incremental regimen of Sustanon

SUMMARY:
"Observational study of clinical outcomes for testosterone treatment of pubertal delay in Duchenne Muscular Dystrophy" is a single centre observational study that aims to follow the progress of 20 adolescents with Duchenne Muscular Dystrophy (DMD) and delayed puberty who are treated by the Newcastle muscle team, as they are treated with testosterone to induce puberty. The participants will all be treated with the standard stepwise regimen of testosterone injections every 4 weeks and data will be collected to help determine the effectiveness and tolerability of the current treatment regimen. The investigators will use the data to explore the effect of testosterone on pubertal development, growth, muscle strength and function, bone mineral density and body composition and characterise any side effects. Semi-structured interviews will also be carried out to learn the boys' views on the tolerability of the regimen. The study will last up to a maximum of 27 months in total for each participant, but may be less if they are happy with pubertal development before this time. It is important to do this study because from the investigator's limited experience in this group, testosterone treatment seems to be well liked and tolerated but the best treatment regimen to use remains unknown and there is no current consensus. It is not currently part of the standard of care in DMD but it would be important to include it if this study can show that it is an effective treatment for pubertal delay.

ELIGIBILITY:
Inclusion Criteria:

* A molecular diagnosis of Duchenne Muscular Dystrophy.
* Males aged between 12 and 17 years of age at time of first dosing
* Prepubertal (Tanner stage 1, testicular volume <4 mls, initial testosterone level of <2.0 nmol/l)
* Subjects are receiving the standard of care for DMD as recommended by the NorthStar UK and TREAT-NMD guidelines
* Patients are capable of sitting upright in a wheelchair for at least an hour
* Patients have stable respiratory function. Artificial ventilation with either Bipap/continuous positive airways pressure (CPAP) or tracheostomy is not a contraindication to the study.
* Informed consent/assent signed by the patient (or parent/guardian if under 16 years of age)

Exclusion Criteria:

* Severe learning difficulties that would preclude them from cooperating with examination.
* Anticipated surgery during the study period.
* Symptomatic cardiac failure.
* Participants/families who may have emotional or psychological problems if recruited to a study
* Hypersensitivity to the active substance or to any of the excipients, including arachis oil or derivatives (including hypersensitivity and allergy to peanuts or soya.)
* Any contra-indication to receiving an intramuscular injection
* Any additional chronic disease that affects androgen production
* Anti-coagulant therapy
* If participation in the study is not recommended in the opinion of the investigators

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a single-centre, prospective, observational, study on clinical outcomes of testosterone replacement therapy in adolescents with DMD and delayed puberty. Being an observational study of routine care, there will be no specified end point. We will aim to recruit any adolescent with DMD and delayed puberty who is reviewed by the muscle team at the John Walton Muscular Dystrophy Research Centre from the study approval date.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Total score in the Treatment Satisfaction Questionnaire for Medication (TSQM) | 2 years

SECONDARY OUTCOMES:
Subject's reported effectiveness of testosterone therapy as assessed by semi-structured interviews pre and post treatment | 2 years
Total score in Northstar Ambulatory Assessment or Performance of the Upper Limb if non-ambulant | 2 years
Z-score from Bone mineral adjusted density of the lumbar spine and total body (minus head) using Dual Xray Absorptiometry (DXA) | 2 years
Percentage of body mass assessed by DXA | 2 years
Osteocalcin level, measured by blood test | 2 years
P1NP level, measured by blood test | 2 years
Percentage fat fraction as assessed by muscle Magnetic Resonance Imaging (MRI) of upper and lower limbs | 2 years
Pubertal staging assessed using Tanner staging and testicular volume | 2 years
Bone age as assessed by wrist and hand X-Ray | 2 years
Hormonal assessment of pubertal staging using testosterone level | 2 years
Forced vital capacity, measured by spirometry | 2 years
Cardiac function, assessed by Electrocardiogram (ECG) and echo | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michela Guglieri, Principal Investigator — Newcastle University
Locations (1):
- Institute of Genetic Medicine, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data available on request

REFERENCES:
- [Derived] Wood CL, Cheetham TD, Hollingsworth KG, Guglieri M, Ailins-Sahun Y, Punniyakodi S, Mayhew A, Straub V. Observational study of clinical outcomes for testosterone treatment of pubertal delay in Duchenne muscular dystrophy. BMC Pediatr. 2019 Apr 25;19(1):131. doi: 10.1186/s12887-019-1503-x. PMID 31023296